CLINICAL TRIAL: NCT04079101
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of BIIB104 in Healthy Japanese and Non-Japanese Participants
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacokinetics of BIIB104 in Healthy Japanese and Non-Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 263HV106
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — PF-04958242

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BIIB104 0.15 mg (Experimental): Participants will receive multiple oral doses of BIIB104 0.15 mg capsules twice daily (BID) for 9 days, with an additional dose occurring in the morning on Day 10.
  Interventions: Drug: BIIB104
- BIIB104 0.5 mg (Experimental): Participants will receive multiple oral doses of BIIB104 0.5 mg capsules BID for 9 days, with an additional dose occurring in the morning on Day 10.
  Interventions: Drug: BIIB104
- Placebo (Experimental): Participants will receive multiple oral doses of placebo-matched BIIB104 capsules BID for 9 days, with an additional dose occurring in the morning on Day 10.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB104 — Administered as specified in the treatment arm.
  Other Names: PF-04958242
  Arms: BIIB104 0.15 mg; BIIB104 0.5 mg
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the pharmacokinetics (PK) of BIIB104 in healthy Japanese and non-Japanese participants. The secondary objective is to evaluate the safety and tolerability of multiple, oral doses of BIIB104 administered BID for 9 days, with an additional dose occurring in the morning on Day 10 in healthy Japanese and non-Japanese participants.

ELIGIBILITY:
Key Inclusion Criteria:

* For Japanese participants, was born in Japan, and biological parents and grandparents were of Japanese origin.
* For Japanese participants, if living outside Japan for more than 5 years, must not have significantly modified diet since leaving Japan.
* Non-Japanese participants must have a screening weight within ±20% of the mean value for Japanese participants.

Key Exclusion Criteria:

* Suicide attempt within the last 2 years. Participants who, in the Investigator's judgment, pose a significant suicide risk or who have suicidal ideation associated with actual intent and a method or plan in the past 6 months (i.e., "Yes" answers on items 4 or 5 of the Columbia Suicide Severity Rating Scale) will be excluded from the study.

Note: Other protocol specific inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 31 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration of BIIB104 | pre-dose on Day 1, 2, 4, 7, 10; 0.25 hour (h), 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 8h and 12h post-dose on Day 1 and 10 ; 1.5h post-dose on Day 4 and 7; Day 11
Time to Reach Maximum Observed Concentration of BIIB104 | pre-dose on Day 1, 2, 4, 7, 10; 0.25 hour (h), 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 8h and 12h post-dose on Day 1 and 10 ; 1.5h post-dose on Day 4 and 7; Day 11
Area Under the Concentration-Time Curve Within a Dosing Interval (AUCtau) of BIIB104 | pre-dose on Day 1, 2, 4, 7, 10; 0.25 hour (h), 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 8h and 12h post-dose on Day 1 and 10 ; 1.5h post-dose on Day 4 and 7; Day 11
Maximum Observed Concentration at Steady State of BIIIB104 | pre-dose on Day 1, 2, 4, 7, 10; 0.25 hour (h), 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 8h and 12h post-dose on Day 1 and 10 ; 1.5h post-dose on Day 4 and 7; Day 11
Time to Reach Maximum Observed Concentration at Steady State of BIIB104 | pre-dose on Day 1, 2, 4, 7, 10; 0.25 hour (h), 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 8h and 12h post-dose on Day 1 and 10 ; 1.5h post-dose on Day 4 and 7; Day 11
Area Under the Concentration-Time Curve Over a Uniform Dosing Interval Tau at Steady State of BIIB104 | pre-dose on Day 1, 2, 4, 7, 10; 0.25 hour (h), 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 8h and 12h post-dose on Day 1 and 10 ; 1.5h post-dose on Day 4 and 7; Day 11
Apparent Total Body Clearance of BIIB104 | pre-dose on Day 1, 2, 4, 7, 10; 0.25 hour (h), 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 8h and 12h post-dose on Day 1 and 10 ; 1.5h post-dose on Day 4 and 7; Day 11
Apparent Volume of Distribution of BIIB104 | pre-dose on Day 1, 2, 4, 7, 10; 0.25 hour (h), 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 8h and 12h post-dose on Day 1 and 10 ; 1.5h post-dose on Day 4 and 7; Day 11
Elimination Half-Life of BIIB104 | pre-dose on Day 1, 2, 4, 7, 10; 0.25 hour (h), 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 8h and 12h post-dose on Day 1 and 10 ; 1.5h post-dose on Day 4 and 7; Day 11
Accumulation Ratio at Steady State of BIIB104 | pre-dose on Day 1, 2, 4, 7, 10; 0.25 hour (h), 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 8h and 12h post-dose on Day 1 and 10 ; 1.5h post-dose on Day 4 and 7; Day 11
Trough Concentration of BIIB104 | pre-dose on Day 1, 2, 4, 7, 10; 0.25 hour (h), 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 8h and 12h post-dose on Day 1 and 10 ; 1.5h post-dose on Day 4 and 7; Day 11

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Baseline (Day 1) up to Day 14
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Number of Participants With Serious Adverse Events (SAEs) | Screening up to Day 14
  An SAE is any untoward medical occurrence that at any dose results in death, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or is a medically important event.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/